CLINICAL TRIAL: NCT01457625
Title: The Association of Serum Fetuin A Level, Insulin Resistance and Hepatic Fat Content and Their Associations With Overall Survival in Maintenance Hemodialysis and Peritoneal Dialysis Patients
Brief Title: Clinical Study of Serum Fetuin A Level, Insulin Resistance and Hepatic Fat Content in Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Yuan Chen, attending physician, Far Eastern Memorial Hospital
Other Study IDs: FEMH - 2011 - C - 006
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Fatty Liver
Keywords: fetuin A liver fat content visceral obesity mortality
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- liver fat contents

SUMMARY:
Background Fetuin A, synthesized in hepatocyte, is a circulatory inhibitor of precipitation of calcium and phosphate and links to cardiovascular calcification and mortality in dialysis patients; besides, it is associated with insulin resistance in general population. Hepatic fat accumulation enhanced fetuin A secretion in animal model.

Objects This study is designed to investigate the association of fetuin A level, insulin resistance and hepatic fat content in dialysis patients. Besides, we planed to observe the survival of dialysis patient with different hepatic fat content.

Methods. This is a prospective observational study. Three hundred and fifty ESRD patients undergoing maintenance HD or PD will be recruited for this prospective investigation. All the participants will receive baseline abdominal ultrasound for estimation of hepatic fat content. Hepatic fat content will be estimated as minimal, mild, moderate or severe according to the Hepburn classification. Besides, all participants also check baseline fetuin A, HOMA-IR, hs-CRP, adiponectin, leptin and lipid profiles (T-CHO, TG, LDL-C, HDL-C), nutritional parameter and other biochemical parameters. All participants will be followed for 4 years for survival analysis. The outcomes are all-cause mortality and composite CV mortality.

Expected results Dialysis patients with higher hepatic fat may have higher fetuin A levels which may lead to long-term survival benefits.

DETAILED DESCRIPTION:
Background:

Fetuin A is a protein secreted by hepatocytes that inhibits insulin receptor tyrosine kinase of adipose and muscle cells (1, 2). Recently, its inhibitory potency on calcium phosphate precipitation has been linked to cardio-vascular (CV) calcification and has predicted CV and non-CV mortality in dialysis patients (3, 4). In most investigations, fetuin A deficiency is associated with higher mortality, worse CV outcomes in dialysis patients. In our recent study, fetuin A deficiency is also linked to vascular access failure in hemodialysis (HD) patients (5). The pathogenesis of worse survival in these fetuin A deficiency dialysis patients is not well-known. Nevertheless, the associations of fetuin A deficiency and progression of vascular calcification and atherosclerosis are thought to be the possible mechanism of the high CV mortality (6, 7).

In general population, fetuin A is associated with insulin resistance, metabolic syndrome and obesity, that is, human with higher fetuin A concentration has higher insulin resistance (8). Insulin resistance, diabetes and metabolic syndrome are all important predictors of long-term CV outcome in general population (9, 10). In an interventional study performed in diabetic human with normal kidney function, treatment with pioglitazone seems to decrease fetuin A levels and enhance insulin sensitivity (11). In an animal model, mice with fatty liver presented up-regulated fetuin A (Ahsg) mRNA expression (1, 2). In non-diabetic subjects, fetuin A is associated with hepatic fat accumulation and insulin resistance (12). Moreover, in a recent investigation, fetuin A concentration was associated with body fat mass in chronic kidney disease (CKD) patients not yet receiving dialysis (13). In our previous investigation, we also found HD patients with higher fetuin A concentration have higher risk to be truncal obesity and hypertriglyceridemia (14). These studies suggested this liver-secreted protein rapidly responds to hepatic fat accumulation which inhibits generation of adiponectin in adipose tissue; therefore higher fetuin-A and lower adiponectin may contribute to obesity-induced insulin resistance and development of diabetes in general population and CKD patients (15). However, this relationship has not been shown in dialysis patients.

Although obesity, metabolic syndrome contributed to higher CV mortality in general population (9, 10); patients under dialysis with higher BMI experienced short-term survival benefit (16). It is so-called "reverse epidemiology" in dialysis patients. Generally speaking, well-nutrition dialysis patients experienced less malnutrition-inflammation complex and therefore, their short-term survival benefit from being well-nutrition overcomes the long-term survival disadvantage brought from over-nutrition such as obesity and insulin resistance. However, ESRD patients with abdominal obesity still have higher CV mortality risk (17).The interesting part of the results these investigations is that, fetuin A deficiency in dialysis patients have worse CV outcome; on the contrary, higher fetuin A level leads to insulin resistance and thereafter higher CV mortality in general population. It is not clear that whether the fetuin A concentration is another "reverse epidemiology" in dialysis patients. But dialysis patients with well-nutrition, presented with higher BMI, more hepatic fat accumulation have better survival. We hypothesize the survival disadvantages of fetuin A deficiency, which is frequently present in dialysis patients, may have a major impact on mortality in a shorter period of time; and increased hepatic fat-accumulation (over-nutrition) may leads to fetuin A secretion and overwhelms the short-term negative effects of fetuin A deficiency on survival, finally, leading to a protective effect of high BMI, hepatic fat accumulation or over-nutrition on overall survival in dialysis patients.

Study purposes:

This study is designed to:

1. To evaluate the association of hepatic fat content and fetuin A concentration in maintenance HD/PD patients
2. To evaluate the association of fetuin A concentration and insulin resistance markers in HD/PD patients
3. To evaluate the overall survival (4-year) of HD/PD patients with different content of hepatic fat

Study designs and methods:

This is a prospective observational study. Three hundred and fifty ESRD patients undergoing maintenance HD or PD for more than 6 months will be recruited for this prospective investigation.

All the participants will receive baseline abdominal ultrasound for estimation of hepatic fat content. Hepatic fat content will be estimated as minimal, mild, moderate or severe according to the Hepburn classification: absent (affecting 0% to 2% of the hepatocytes), minimal (2% to 10%), mild (10% to 30%), moderate (30% to 60%), and severe (more than 60% of the hepatocytes). We choose abdominal ultrasound as the method of hepatic fat estimation rather than MRI and CT which are the gold standard of hepatic fat estimation, because the limited use of MRI in dialysis patients and increased cancer risk receiving screening CT. Besides, all participants also check baseline fetuin A, HOMA-IR, hs-CRP, adiponectin, leptin and lipid profiles (T-CHO, TG, LDL-C, HDL-C), nutritional parameter and other biochemical parameters. All participants will be followed for 4 years for survival analysis. The outcomes are all-cause mortality and composite CV mortality.

ELIGIBILITY:
Inclusion Criteria:

1. ESRD patients undergoing maintenance HD or PD for more than 6 months
2. Age>20

Exclusion Criteria:

1. Recent hospitalization duet active medical or psychiatric problems
2. Active malignancy
3. Patient refusal

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three hundred and fifty ESRD patients undergoing maintenance HD or PD will be recruited for this prospective investigation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
liver fat contents, fetuin A levels | 1 year

SECONDARY OUTCOMES:
CV and all-cause mortality | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yuan Chen, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (2):
- Taiwan (2):
  - Far Eastern Memorial Hospital, New Taipei City
  - Far eastern memorial hospital, New Taipei City

REFERENCES:
- [Derived] Chen HY, Tsai WC, Chiu YL, Hsu SP, Pai MF, Yang JY, Peng YS. Triglyceride to high-density lipoprotein cholesterol ratio predicts cardiovascular outcomes in prevalent dialysis patients. Medicine (Baltimore). 2015 Mar;94(10):e619. doi: 10.1097/MD.0000000000000619. PMID 25761189
- [Derived] Chen HY, Chiu YL, Chuang YF, Hsu SP, Pai MF, Yang JY, Peng YS. Visceral adiposity index and risks of cardiovascular events and mortality in prevalent hemodialysis patients. Cardiovasc Diabetol. 2014 Oct 4;13:136. doi: 10.1186/s12933-014-0136-5. PMID 25280960